CLINICAL TRIAL: NCT00260871
Title: Genetic Epidemiological Study of Lung Cancer in Taiwan and Clinical Applications-focusing on Female Lung Adenocarcinoma (GEFLAC)
Brief Title: Genetic Epidemiological Study of Lung Cancer in Taiwan and Clinical Applications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University (Other)
Responsible Party: Dr. Chao Agnes Hsiung, Institute of Population Health Sciences, National Health Research Instiutes, Taiwan
Other Study IDs: 94LCP005; 1.DOH-94-TD-G-111-025; 2.DOH-94-TD-G-111-027
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Lung Cancer
Keywords: lung adenocarcinoma; genetic epidemiology; environmental factors; genetic map; coordination center
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Lung adenocarcinoma in Chinese females is hypothesized to be determined by both genetic and environmental factors. In this grant proposal, we propose to map the loci of susceptibility genes of female lung adenocarcinoma based on multiplex families recruited in Taiwan. We focus on a unique pathological type of a unique population in order to reduce heterogeneity of the genetic background. Compared with western women, female Chinese population has a high prevalence of lung adenocarcinoma. Our reasoning is that if we focus on a specific sub-type, which has a familial basis, we will increase the probability of identifying genes associated with female lung adenocarcinoma. The primary goal of this study is to identify the genetic and environmental determinants of female lung adenocarcinoma, and study the relationship between gene polymorphisms and clinical manifestation profiling of lung cancer.

DETAILED DESCRIPTION:
This research proposal intends to integrate epidemiologists, biostatisticians, clinicians, molecular biologists/geneticists to identify susceptible genes for lung cancer, especially for female lung adenocarcinoma, and to study the relationship between gene polymorphisms and clinical outcomes of lung cancer patients. Our objective is to find gene markers for developing useful screening tools for the high risk group in order to prevent or early detect lung cancer, especially female lung adenocarcinoma.

The specific aims of this subproject include:

1. Establish and maintain the research network that will recruit and follow up the subjects and families for the GEFLAC study; keeping control of the progress of the study.
2. Coordinate all the subprojects such as integrating genotyping data with clinical data and environment data.
3. Continue to employ the candidate gene approach to examine the contribution of specific genes to the lung cancer.
4. Generate genotyping data for candidate genes in the exploring stage and prioritize SNPs of candidate genes for large scale studies.
5. Identify susceptible genes/candidate genes to develop multiplex PCR for screening.

ELIGIBILITY:
Inclusion Criteria:

* lung adenocarcinoma

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The program project intend to identify susceptible genes for lung cancer, especially for female lung adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsiung, PhD, Study Director — NHRI
Locations (1):
- Division of Biostatistics and Bioinformatics, NHRI, Miaoli County, Taiwan

REFERENCES:
- See also: Related Info — http://www.nhri.org.tw